CLINICAL TRIAL: NCT02983331
Title: Patients With Mortality After Endoscopic Retrograde Cholangiopancreatography
Brief Title: Mortality After Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Type: Observational
Sponsor: Gulsah Karaoren (Other Government)
Responsible Party: Sponsor-Investigator, Gulsah Karaoren, MD, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: GK11
Record Dates: First submitted 2016-11-27; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Mortality; Deep Sedation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: complications during procedure — patients may have anesthesia related complications during procedure

SUMMARY:
In this study, the investigators aimed to overview patients with specific and non-specific complications who admitted to intensive care unit following endoscopic retrograde cholangiopancreatography and had fatal course in the facility

DETAILED DESCRIPTION:
The investigators retrospectively reviewed patients who underwent elective or emergent endoscopic retrograde cholangiopancreatography at semi-prone position under pharyngeal anesthesia (lidocaine spray) with routine monitoring (including electrocardiography, non-invasive blood pressure, peripheral capillary oxygen saturation) and standard sedation protocol (midazolam 0.02 mgkg-1; fentanyl, 1 mgkg-1; propofol 1 mgkg-1) between 2011 and 2016 after approval of local ethics committee of Umraniye Training Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective or emergent ERCP at semi-prone position with routine monitoring and standard sedation protocol

Exclusion Criteria:

* Patients who discharged to ward after treatment and follow-up in ICU

Ages: 42 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively reviewed 1471 patients who underwent elective or emergent ERCP at semi-prone position under pharyngeal anesthesia (lidocaine spray) with routine monitoring (including electrocardiography, non-invasive blood pressure, peripheral capillary oxygen saturation) and standard sedation protocol
Sampling Method: Non-Probability Sample
Enrollment: 1471 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With endoscopic retrograde cholangiopancreatography Related complications | 5 years
  We retrospectively reviewed patients who underwent elective or emergent endoscopic retrograde cholangiopancreatography at semi-prone position under pharyngeal anesthesia (lidocaine spray) with routine monitoring (including electrocardiography, non-invasive blood pressure, peripheral capillary oxygen saturation) and standard sedation protocol
Rate of anaesthesia related mortality of the endoscopic retrograde cholangiopancreatographyprocedure under sedation | 5 years
  We identified patients who developed complications during procedure and admitted to intensive care unit (ICU).

SECONDARY OUTCOMES:
Value of Acute Physiology and Chronic Health Evaluation (APACHE II) score for predicting mortality | 5 years
Value of Charlson comorbidity index (CCI) score for predicting mortality | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gulsah Karaoren, MD, Principal Investigator — Umraniye Research Hospital
Locations (1):
- Istanbul Umraniye Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Katsinelos P, Lazaraki G, Chatzimavroudis G, Gkagkalis S, Vasiliadis I, Papaeuthimiou A, Terzoudis S, Pilpilidis I, Zavos C, Kountouras J. Risk factors for therapeutic ERCP-related complications: an analysis of 2,715 cases performed by a single endoscopist. Ann Gastroenterol. 2014;27(1):65-72. PMID 24714755